CLINICAL TRIAL: NCT01914991
Title: Treatment of the PIP Joint Flexion Contracture: Combined Static and Dynamic Orthotic Intervention Compared With Traditional Combine Therapy. A Randomized Controlled Trial
Brief Title: Combined Static and Dynamic Orthotic Treatment of the PIP Joint
Acronym: StaDinOrt
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FCCSS-UMA-02-13
Record Dates: First submitted 2013-07-24; First posted 2013-08-02 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Health Behaviour
Keywords: proximal interphalangeal joint; Orthoses
MeSH Terms: interventions — Orthotic Devices; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): Conventional treatment: The treatment consisted of 10 minutes of local thermotherapy (paraffin), active exercises at the PIPJ and DIPJ (Distal interphalangeal joint), 3 sets of 15 repetitions of each exercise extending and flexing of the PIPJ with metacarpophalangeal joint from 0° to 90° respectively. Distal interphalangeal joint exercises were conducted with identical repetitions. The metacarpophalangeal joint and PIPJ exercises took place at 0 ° and involved stretching (5 sets of 3 reps, holding for 10 seconds) and Therapeutic U.S (0.8 w/cm2 / 7 minutes).
  Interventions: Procedure: conventional treatment Physical Therapy
- Experimental group (Experimental): dynamic extension contracture orthotic. A mobilizing force of 250 - 300 gm/cm2 was set in each one. Patients were instructed to wear it for at least 6 hours per day and then removed it for ADL (Activity Daily Living). A static orthosis was constructed using orfitcast material to the maximum, pain-free length allowed by the tissues at night. Static and dynamic orthoses were checked once a week and adjusted as necessary.
  Interventions: Procedure: dynamic extension contracture orthotic

INTERVENTIONS:
Procedure: dynamic extension contracture orthotic — A dynamic orthosis was constructed in the experimental group using the same style of dynamic extension contracture orthotic. A mobilizing force of 250 - 300 gm/cm2 was set in each one. Patients were instructed to wear it for at least 6 hours per day and then removed it for ADL (Activity Daily Living). A static orthosis was constructed using orfitcast material to the maximum, pain-free length allowed by the tissues at night. Static and dynamic orthoses were checked once a week and adjusted as necessary.
  Other Names: ORTHOTIC
  Arms: Experimental group
Procedure: conventional treatment Physical Therapy — Traditional treatment was applied to one control group. The treatment consisted of 10 minutes of local thermotherapy (paraffin), active exercises at the PIPJ and DIPJ (Distal interphalangeal joint), 3 sets of 15 repetitions of each exercise extending and flexing of the PIPJ with metacarpophalangeal joint from 0° to 90° respectively. Distal interphalangeal joint exercises were conducted with identical repetitions. The metacarpophalangeal joint and PIPJ exercises took place at 0 ° and involved stretching (5 sets of 3 reps, holding for 10 seconds) and Therapeutic U.S (0.8 w/cm2 / 7 minutes).
  Other Names: PHYSICAL THERAPY
  Arms: Control group

SUMMARY:
Study Design: Randomized controlled clinical study. Introduction: Physiotherapeutic intervention aiming to restore mobility using different techniques as stretching, hot packs, exercises, therapeutic ultrasound and orthotics. No scientific evidence has been found correlating improved joint mobility and the use of these techniques. Application techniques of orthoses to reshape the soft tissues have been well detailed, however, no scientific evidence supporting their effectiveness on proximal interphalangeal joint (PIPJ) lag extension resolution using them as a single treatment has been found.

Purpose of the Study: The purpose of the study was to test the effectiveness of static and dynamic orthosis in patients with a PIPJ flexion retraction using them as a single treatment compared with traditional combined therapies.

Method: 63 participants were included in the study. Patients who used splints were compared to a control group who received conventional treatment. Active and passive mobility were measured before the experiment and again three months after. All the patients were measured under the same conditions and treated by the same hand therapist. The relationship between contracture resolution and function was measured using the DASH Spanish Version.

ELIGIBILITY:
INCLUSION CRITERIO:

* 18 years old
* had given their consent
* having suffered trauma to the hand or finger which has resulted in joint damage with a consequent loss of full extension of the PIPJ
* duration of the injury being between four and 30 weeks.

EXCLUSION CRITERIA:

* Patients who had no proper joint alignment,
* Patients those with a presence of nerve or tendon associated dupuytren,
* campodactilea
* tubular bone fractures
* acute inflammatory signs
* joint instability
* avascular necrosis
* infection of the affected finger were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Active Range of motion AROM (degrees) | baseline; post-treatment (3 moths)
  AROM and function were measured in all patients at inclusion and at three months after the start of the study. which was measured using a short arm goniometer Stainless Baseline 180°. A lateral measurement following the standardized protocol recommended by the American Society of Hand Therapists was used.

SECONDARY OUTCOMES:
Disability of the arm shoulder AND HAND (DASH QUESTIONNAIRE) | baseline; post-treatment (3 moths); 24 weeks follow up
  The Spanish standard version of DASH instrument (Rosales et al. 2002) (www.dash.iwh.on.ca) for measuring upper extremity disability was used as a secondary outcome measurement. The questionnaire was given to the participants the day before starting the treatment and again after three months.
changes from postreatment Active range of Motion (AROM) degrees | 24 weeks follow up
  AROM and function were measured in all patients at inclusion and at three months after the start of the study. which was measured using a short arm goniometer Stainless Baseline 180°. A lateral measurement following the standardized protocol recommended by the American Society of Hand Therapists was used.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, PhD, Study Director — University of Malaga
Locations (1):
- Centro Tecan, Málaga, Malaga, Spain

REFERENCES:
- [Derived] Cantero-Tellez R, Cuesta-Vargas AI, Cuadros-Romero M. Treatment of proximal interphalangeal joint flexion contracture: combined static and dynamic orthotic intervention compared with other therapy intervention: a randomized controlled trial. J Hand Surg Am. 2015 May;40(5):951-5. doi: 10.1016/j.jhsa.2015.01.005. Epub 2015 Mar 11. PMID 25771480